CLINICAL TRIAL: NCT02991040
Title: A Multicenter, Double-Blind, Randomized, Split-Face Study to Evaluate the Safety and Efficacy of Revanesse® Ultra + (With Lidocaine) Versus Revanesse® Ultra for the Correction of Nasolabial Folds (NLF)
Brief Title: Study to Evaluate Safety and Efficacy of Revanesse® Ultra + vs Revanesse® Ultra for Correction of NLF
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Prollenium Medical Technologies Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: SYM2016-02
Record Dates: First submitted 2016-12-06; First posted 2016-12-13 (Estimated); Results first posted 2019-04-11 (Actual); Last update posted 2019-04-11 (Actual); Status verified 2019-03

CONDITIONS: Nasolabial Fold Correction

STUDY DESIGN:
Intervention Model Description: Subjects were treated with Revanesse Ultra in the NLF on one side of the face and Revanesse Ultra+ in the NLF on the other side of the face. The side of the face for each study product was randomly assigned.
Who Masked: Outcomes Assessor
Masking Description: The side of the face for each product was randomly assigned. The investigator performing the evaluations and the subject were blinded to the treatment; injections of the study product were performed by an unblinded injecting investigator.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Device: Yes

ARMS (1):
- Revanesse Ultra+ (Experimental): Revanesse Ultra+ (with lidocaine) vs Revanesse Ultra without lidocaine
  Interventions: Device: Revanesse Ultra+ (with lidocaine); Device: Revanesse Ultra

INTERVENTIONS:
Device: Revanesse Ultra+ (with lidocaine) — Bilateral nasolabial fold trial to compare the safety and efficacy profiles of Revanesse® Ultra + (with lidocaine) to Revanesse® Ultra (comparator)
  Other Names: Revanesse Versa+
Device: Revanesse Ultra — Comparator without lidocaine
  Other Names: Revanesse Versa

SUMMARY:
A Multicenter, Double-Blind, Randomized, Split-Face Study to Evaluate the Safety and Efficacy of Revanesse® Ultra + (with Lidocaine) versus Revanesse® Ultra for the Correction of Nasolabial Folds to compare the safety and efficacy profiles of Revanesse® Ultra + (with lidocaine, hereafter referred to as Revanesse Ultra +) to Revanesse Ultra for subjects undergoing correction of nasolabial folds (NLFs)

DETAILED DESCRIPTION:
This is a randomized, multicenter, double-blind, split-face study in subjects seeking nasolabial fold correction. Subjects will be treated with Revanesse Ultra + in the NLF on one side of the face and Revanesse Ultra in the NLF on the other side of the face. The side of the face for each study product will be randomly assigned. The investigator and the subject will be blinded to the treatment; injections of the study product will be performed by an unblinded injecting investigator.

At each visit, investigator and subject evaluations of the treated areas will be performed and recorded

ELIGIBILITY:
Inclusion Criteria:

* Subjects must meet all of the following criteria to be eligible for the study:

  1. Men or women 22 years of age or older seeking augmentation therapy for correction of bilateral nasolabial folds.
  2. Two fully visible bilateral nasolabial folds each with a Wrinkle Severity Rating Scale Score (WSRS) of 3 or 4 that may be corrected with an injectable dermal filler. The NLFs should be symmetrical, i.e., WSRS scores at NLFs on both sides should be the same (both Moderate [3] or both Severe [4]).
  3. If female and of childbearing potential, a negative urine pregnancy test and agree to use adequate contraception. Female subjects of childbearing potential (excluding women who are surgically sterilized or postmenopausal for at least 2 years) must have a negative urine pregnancy test and must be willing to use a medically accepted method of contraception during the study. The following are considered acceptable methods of birth control for the purpose of this study: oral contraceptives, contraceptive patches, contraceptive implant, vaginal contraceptive, double barrier methods (e.g., condom and spermicide), contraceptive injection (Depo-Provera®), intrauterine device (IUD), hormonal IUD (Mirena®), and abstinence with a documented second acceptable method of birth control if the subject becomes sexually active. Subjects entering the study who are on hormonal contraceptives must have been on the method for at least 90 days prior to the study and continue the method for the duration of the study. Subjects who had used hormonal contraception and stopped must have stopped no less than 90 days prior to Visit 1/Day 1.
  4. Ability to understand and comply with the requirements of the study.
  5. Willingness and ability to provide written informed consent. 6. Agree to refrain from seeking other treatment for this condition during the study.

Exclusion Criteria:

Subjects who meet any of the following criteria will be excluded from the study:

1. Wrinkle Severity Rating Scale Score of ≤ 2 on the right or left nasolabial fold.
2. Women who are pregnant or lactating.
3. Received prior dermabrasion, facelift, or Botox below the orbital rim, or had undergone procedures based on active dermal response (e.g., laser or chemical peeling procedures) within 6 months (180 days) prior to study entry.
4. Use of any facial tissue augmenting therapy with non-permanent filler or aesthetic facial surgical therapy within 9 months prior to study entry.
5. Has ever received semi-permanent fillers anywhere in the face or neck, or is planning to be implanted with these products during the study.
6. Has a permanent implant placed in the NLF area.
7. Evidence of scar-related disease or delayed healing activity within the past 1 year.
8. Scars at the intended treatment sites.
9. History of keloid formation or hypertrophic scars.
10. Any infection or unhealed wound on the face.
11. Allergic history including anaphylaxis, multiple severe allergies, atopy, or allergies to natural rubber latex, lidocaine or any amide-based anesthetic, hyaluronic acid products, or Streptococcal proteins or have plans to undergo desensitization therapy during the term of the study.
12. Aspirin or nonsteroidal anti-inflammatory drugs within 1 week (7 days) prior to treatment.
13. Concomitant anticoagulant therapy, antiplatelet therapy, or history of bleeding disorders, coagulation defects or connective tissue disorders.
14. Over-the-counter (OTC) wrinkle products or prescription wrinkle treatments within 4 weeks (28 days) prior to treatment and throughout the study.
15. Immunocompromised or immunosuppressed.
16. Clinically significant organic disease including clinically significant cardiovascular, hepatic, pulmonary, neurologic, or renal disease or other medical condition, serious intercurrent illness, or extenuating circumstance that, in the opinion of the investigator, preclude participation in the trial.
17. Received any investigational product within 30 days of signing the Informed Consent Form.
18. Facial tattoo that may interfere with diagnosis.
19. Systemic (oral/injectable) corticosteroids or immunosuppressive medications within 30 days prior to treatment and topical steroids on the face within 14 days prior to treatment start and throughout the study.
20. Acne and/or other inflammatory diseases of the skin.
21. Acute or chronic skin disease, inflammation or related conditions, cancerous or precancerous lesions on or near the injection sites.-

Min Age: 22 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2016-08 (Actual); Primary Completion 2017-08 (Actual); Study Completion 2017-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael H. Gold, MD, Principal Investigator — Tennessee Clinical Research, Inc
Locations (1):
- Tennessee Clinical Research Center, Nashville, Tennessee, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was undertaken between August 24 2016 and June 21 2017. Subjects that were randomized, there were 100 intent-to-treat (ITT), 95 modified intent-to-treat (mITT), 75 per-protocol (PP) subjects. Of the subjects randomized there were 17 subjects in the rollover subset (17 ITT, 12 mITT, and 12 PP subjects).
  96 Subjects completed the study.
Groups:
- Revanesse Ultra+: Revanesse Ultra+ (with lidocaine)
  Revanesse Ultra+ (with lidocaine): Bilateral nasolabial fold trial to compare the safety and efficacy profiles of Revanesse® Ultra + (with lidocaine) to Revanesse® Ultra (comparator)
  Revanesse Ultra: Comparator without lidocaine
Period: Overall Study
Arm/Group | Revanesse Ultra+
Started | 100
Completed | 96
Not Completed | 4
Not completed — Withdrawal by Subject | 2
Not completed — Lost to Follow-up | 2

BASELINE CHARACTERISTICS:
Population: There were 100 subjects randomized, in accordance with the inclusion / exclusion criteria, who were men or women at least 22 years of age with two fully visible bilateral nasolabial folds each with a Wrinkle Severity Rating Scale (WSRS) score of 3 or 4 (moderate or severe)
Arm/Group | Revanesse Ultra+
Number analyzed (Participants) | 100
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | NA — exclusion criteria
  Between 18 and 65 years | 73
  >=65 years | 21
Age, Continuous [Mean (Full Range); unit: years] | 58.0 [30 to 83]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 93
  Male | 7
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 38
  Not Hispanic or Latino | 62
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 10
  White | 89
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 100

OUTCOME MEASURES:

1. Primary Outcome: Pain at Injection as Measured by Subject on a 100 mm Visual Analog Scale (VAS) Scale at Time 0 Minutes Post Injection
Description: Visual Analog Scale for Pain. A 100 mm scale with 0 mm being no pain (best outcome) to 100 mm being worst pain (worst outcome). The higher scores mean a worse outcome
Time Frame: at injection Time 0
Population: mITT: All randomized subjects who met the inclusion/exclusion criteria, were randomized, received both study products, and had VAS pain score immediately post injection from both sides of the face
Measure: Mean (Standard Deviation); unit: VAS
Groups:
- Revanesse Ultra: Revanesse Ultra (without lidocaine)
Arm/Group | Revanesse Ultra+ | Revanesse Ultra
Number analyzed (Participants) | 95 | 95
VAS | 26.2 (24.51) | 39.4 (25.45)

2. Secondary Outcome: Pain Measured by Subject on 100 mm VAS Scale at 15, 30, 45, and 60 Minutes Post Injection and at 2 Weeks Post Injection
Description: Visual Analog Scale for pain. A 100 mm scale with 0 mm being no pain (best outcome) to 100 mm being worst pain (worst outcome). The higher score means a worse outcome.
Time Frame: 15, 30, 45, and 60 minutes post injection and at 2 weeks post injection
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: VAS score
Arm/Group | Revanesse Ultra+ | Revanesse Ultra
Number analyzed (Participants) | 95 | 95
VAS score
  15 minutes post injection | 9.52 (14.83) | 15.26 (18.37)
  30 minutes post injection | 4.72 (9.10) | 7.46 (11.06)
  45 minutes post injection | 2.66 (6.61) | 4.21 (7.89)
  60 minutes post injection | 2.13 (6.39) | 2.86 (7.28)
  2 weeks post injection | 0.25 (1.07) | 0.25 (1.07)

3. Secondary Outcome: Wrinkle Severity Rating Score (WSRS)
Description: The Wrinkle Severity Rating Scale is a 5-point scale with 1 = Absent; 2 = Mild; 3 = Moderate; 4 = Severe and 5 = Extreme. 1 is the best outcome while 5 is the worst outcome. The higher scores mean a worse outcome.
Time Frame: Visit 2/Day 14 (± 2 days), Visit 3/Day 28 (± 2 days), Visit 4/Day 84 (± 4 days), Visit 5/Day 168 (Week 24) (± 7 days)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Wrinkle Severity Rating scale
Arm/Group | Revanesse Ultra+
Number analyzed (Participants) | 95
Wrinkle Severity Rating scale
  Visit 2/Week 2 | -0.03 (0.402)
  Visit 3/ Week 4 | 0.02 (0.25)
  Visit 4/Week 12 | 0.00 (0.21)
  Visit 5/Week 24 | -0.02 (0.25)

4. Secondary Outcome: Patient Global Aesthetic Improvement
Description: Patient Global Aesthetic Improvement Score is a 5-point scale used to assess the subject's satisfaction with the visual appearance of their NLF correction after treatment. 1 = Worse (worst outcome), 2 = No Change, 3 = Improved, 4 = Much Improved, 5 = Very Much improved (best outcome). The higher scores mean a better outcome.
Time Frame: Visit 2/Day 14 (± 2 days), Visit 3/Day 28 (± 2 days), Visit 4/Day 84 (± 4 days), Visit 5/Day 168 (Week 24) (± 7 days)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Revanesse Ultra+
Number analyzed (Participants) | 93
score on a scale
  Visit 2/Week 2 | 0.04 (.35)
  Visit 3/Week 4 | -0.10 (0.42)
  Visit 4/Week 12 | -0.07 (0.38)
  Visit 5/Week 24 | 0.00 (0.46)

5. Secondary Outcome: Investigator Global Aesthetic Improvement
Description: Investigator Global Aesthetic Improvement Score is a 5-point scale with 1 = Worse (worst outcome); 2 = No Change; 3 = Improved; 4 = Much Improved, 5 = Very much improved (best outcome). The higher scores mean a better outcome.
Time Frame: Visit 2/Day 14 (± 2 days), Visit 3/Day 28 (± 2 days), Visit 4/Day 84 (± 4 days), Visit 5/Day 168 (Week 24) (± 7 days)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Revanesse Ultra+
Number analyzed (Participants) | 93
score on a scale
  Visit 2/Week 2 | 0.02 (0.48)
  Visit 3/Week 4 | -0.02 (0.14)
  Visit 4/Week 12 | -0.01 (0.18)
  Visit 5/Week 24 | 0.03 (0.17)

6. Other Pre Specified Outcome: Safety and Tolerability of Revanesse Ultra and Revanesse Ultra+ Injection by Incidence of Treatment Emergent Adverse Events
Description: study products will be compared by evaluating the nature, severity, and frequency of treatment-emergent adverse events (TEAEs)
Time Frame: at injection, Visit 2/Day 14 (± 2 days), Visit 3/Day 28 (± 2 days), Visit 4/Day 84 (± 4 days), Visit 5/Day 168 (Week 24) (± 7 days)
Population: ITT (safety population): All randomized subjects who received study product
Measure: Number; unit: events
Arm/Group | Revanesse Ultra+ | Revanesse Ultra
Number analyzed (Participants) | 100 | 100
events | 112 | 102

ADVERSE EVENTS:
Time Frame: Each subject was monitored for the occurrence of AEs, including SAEs, immediately after treatment initiation. Each subject was followed for safety monitoring until discharged from the study. Follow-up procedures related to pregnancy or AEs or SAEs could continue beyond the end of the study. Adverse event data was collected over a 10 month period of time.
Arm/Group | Revanesse Ultra+ | Revanesse Ultra
All-Cause Mortality (participants affected / at risk) | 0/100 | 0/100
Serious Adverse Events (participants affected / at risk) | 0/100 | 1/100
Other Adverse Events (participants affected / at risk) | 53/100 | 52/100
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Revanesse Ultra+ (N=100) | Revanesse Ultra (N=100)
Worsening Right Knee Pain (arthralgia) (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Revanesse Ultra+ (N=100) | Revanesse Ultra (N=100)
Injection Site Bruising (General disorders) | 32 (37) | 31 (39)
Injection site pain (General disorders) | 17 (19) | 21 (28)
Injection site swelling (General disorders) | 21 (23) | 17 (21)
Injection site erythema (General disorders) | 15 (17) | 12 (13)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2016-07-08): https://cdn.clinicaltrials.gov/large-docs/40/NCT02991040/Prot_000.pdf
  • Statistical Analysis Plan (2017-07-21): https://cdn.clinicaltrials.gov/large-docs/40/NCT02991040/SAP_001.pdf